CLINICAL TRIAL: NCT00426283
Title: A Double Blinded, Randomized Trial of Swallowed 1760mcg Fluticasone Propionate Versus Placebo in the Treatment of Eosinophilic Esophagitis
Brief Title: A Study of Flovent in Patients With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marc Rothenberg, MD (Other)
Responsible Party: Sponsor-Investigator, Marc Rothenberg, MD, Marc Rothenberg, MD, PhD, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-10-07
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flovent 1760 mcg (Experimental): Fluticasone propionate 880 mcg twice daily for 3 months
  Interventions: Drug: Flovent
- Placebo (Placebo Comparator): Placebo twice daily for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Flovent — 1760 mcg daily
  Other Names: Fluticasone propionate
  Arms: Flovent 1760 mcg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effects (both good and bad) of high dose swallowed fluticasone propionate (Flovent) in subjects with eosinophilic esophagitis (EoE).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for study by subject, or parent/guardian if subject is a minor. Assent will be obtained from all minors 11 years of age and older.
* Histological findings on esophageal biopsy to include peak eosinophil density ≥ 24 per high power field (400x) in the proximal or distal esophagus validated by a pathologist at CCHMC.
* Allergy evaluation including skin-prick testing with multiple food antigens to ensure elimination diet is not indicated.
* Have undergone a minimum 3 months of elimination diet as indicated by skin-prick testing without detectable resolution by repeat endoscopy with biopsies demonstrating persistent EE OR subject/parental refusal to follow elimination diet. If the subject/parent refuses the elimination diet, they are eligible for this study.
* Treatment with a proton-pump inhibitor for at least two months (rounded to nearest month) prior to endoscopy OR failure of histological improvement as defined by < 1 eosinophil per HPF after 2 month (rounded to nearest month) trial of proton pump inhibitor documented by prior endoscopy. The PPI must be used prior to endoscopy to rule out the possibility of GERD.

Exclusion Criteria:

* History of poor tolerance to Fluticasone Propionate (FP), as defined as multiple episodes of oral candidiasis, hypothalamic-pituitary-adrenal axis suppression as evidenced by signs of Cushing syndrome, headaches, or increased respiratory infections during exposure to Flovent
* Unable to cooperate with use of MDI
* Pregnant females
* Concurrent or recent (within 3 months) use of systemic corticosteroids.
* Unable to swallow medicines (i.e., fed only by gastrostomy tube).
* Comorbid eosinophilic disorders.
* Previously treated with swallowed glucocorticoid for EE within 3 months of the screening visit. Nasal glucocorticoids taken for EE are permitted.

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, M.D., Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - The Children's Hospital of Denver, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Butz BK, Wen T, Gleich GJ, Furuta GT, Spergel J, King E, Kramer RE, Collins MH, Stucke E, Mangeot C, Jackson WD, O'Gorman M, Abonia JP, Pentiuk S, Putnam PE, Rothenberg ME. Efficacy, dose reduction, and resistance to high-dose fluticasone in patients with eosinophilic esophagitis. Gastroenterology. 2014 Aug;147(2):324-33.e5. doi: 10.1053/j.gastro.2014.04.019. Epub 2014 Apr 22. PMID 24768678
- See also: Cincinnati Center for Eosinophilic Disorders — http://www.cchmc.org/cced

RESULTS

PARTICIPANT FLOW:
Groups:
- Flovent 1760 mcg: Drug
  Flovent : 1760 mcg daily
- Placebo: Placebo twice daily
Period: Overall Study
Arm/Group | Flovent 1760 mcg | Placebo
Started | 28 | 14
Completed | 23 | 13
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Flovent 1760 mcg: Drug
  Flovent : 880 mcg twice daily
- Total: Total of all reporting groups
Arm/Group | Flovent 1760 mcg | Placebo | Total
Number analyzed (Participants) | 28 | 14 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 12 | 38
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.15 (6.42) | 13.54 (7.11) | 12.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 22 | 13 | 35
Region of Enrollment [Number; unit: participants]
  United States | 28 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Attained Remission.
Description: Remission is considered achieved when the highest eosinophil count per high power field (hpf) in all esophageal biopsies is </= 1 eosinophil/hpf after 3 months of therapy.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flovent 1760 mcg | Placebo
Number analyzed (Participants) | 23 | 13
percentage of participants | 65.2 [44.9 to 81.2] | 0 [0 to 22.8]

2. Secondary Outcome: Percent of Participants With Decreased Cortisol Levels After 3 Months
Description: Blood and saliva cortisol was measured and compared to reference range at 3 months. Participants with measures below the reference range were considered "decreased".
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Flovent 1760 mcg | Placebo
Number analyzed (Participants) | 23 | 13
percentage of participants | 17.4 | 0

3. Secondary Outcome: Association of Subject Age, Body Mass Index Z-score, and Allergic Status to Response to Flovent
Description: Strength of the association (odds ratio) of age, body mass index (BMI) z-score , and allergic status with response to Flovent. Allergic status is defined as a history of allergic disease (allergic rhinitis, hay fever, atopic dermatitis, eczema, food anaphylaxis, asthma, or positive skin prick tests). Response is defined as <= 1 eosinophil/high power field in esophageal biopsies.
Time Frame: 3 months
Population: Analysis population is restricted only to those that were given Flovent for the purpose of determining whether these specific variables are associated with response to drug
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Flovent 1760 mcg
Number analyzed (Participants) | 23
Odds Ratio
  Odds Ratio for Age | 0.907 [0.779 to 1.055]
  Odds Ratio for BMI Z-Score | 0.541 [0.205 to 1.433]
  Odds Ratio for Allergic Status | 0.572 [0.049 to 6.607]

4. Secondary Outcome: EoE Score After 3 Months
Description: The gene expression profile is associated with an EoE score algorithm reflecting disease status and severity in a quantifiable number - called the EoE score, based on a core set of 77 diagnostic genes. The EoE score was calculated for Flovent responders and placebo. Higher scores indicate normalization of genes associated with inflammation and fibrosis (disease severity). Therefore higher scores mean a better outcome. The minimum score is zero. There is no maximum score.
Time Frame: 3 months
Population: Population includes only responders to Flovent and all participants finishing the study on Placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Flovent 1760 mcg Responders: Drug
  Flovent : 1760 mcg daily
Arm/Group | Flovent 1760 mcg Responders | Placebo
Number analyzed (Participants) | 15 | 13
score on a scale | 382 (47) | 152 (119)

5. Secondary Outcome: Association of Compliance With Therapy and Response to Flovent
Description: Odds ratio was determined to show the strength of the association between compliance with the drug therapy and response to the drug therapy
Time Frame: 3 months
Population: Analysis population is restricted only to those that were given Flovent for the purpose of determining whether compliance with therapy was associated with response to drug
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Flovent 1760 mcg
Number analyzed (Participants) | 23
Odds Ratio | 1.037 [0.988 to 1.089]

6. Secondary Outcome: Percent of Participants With Abdominal Pain After Therapy
Description: Percent of participants responding that they experienced abdominal pain (i.e. they did not respond "never") after therapy. Responses were dichotomized into "Never" and "sometimes".
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Flovent 1760 mcg | Placebo
Number analyzed (Participants) | 23 | 12
percentage of participants | 63 | 50

ADVERSE EVENTS:
Time Frame: From consent to cessation of treatment which was approximately 4 months
Description: Adverse events were reported according to the MedDRA System Organ Class
Groups:
- Placebo: Placebo : daily
Arm/Group | Flovent 1760 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/14
Other Adverse Events (participants affected / at risk) | 19/28 | 9/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flovent 1760 mcg (N=28) | Placebo (N=14)
General Disorders (General disorders) | 1 (1) | 1 (1)
General Disorders (Eye disorders) | 0 (0) | 2 (2)
General Disorders (Gastrointestinal disorders) | 7 (10) | 2 (2)
General Disorders (Immune system disorders) | 2 (3) | 0 (0)
General Disorders (Infections and infestations) | 3 (4) | 3 (3)
General Disorders (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
General Disorders (Investigations) | 5 (5) | 1 (4)
General Disorders (Nervous system disorders) | 4 (5) | 0 (0)
General Disorders (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (3)
General Disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No